CLINICAL TRIAL: NCT05995132
Title: Compromised Sleep and Circadian Health After Critical Illness: From Diagnosis to Prediction (CHRONOCRIT)
Acronym: CHRONOCRIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut de Recerca Biomèdica de Lleida (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Adriano Targa, PhD, Institut de Recerca Biomèdica de Lleida
Other Study IDs: PI22/00216
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Circadian Dysregulation; Sleep Fragmentation
Keywords: microRNA; circadian rhythms; intensive care unit; sleep; critical survivors
MeSH Terms: conditions — Chronobiology Disorders; Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * 2 Tubes EDTA (6ml)
  * 1 tempus RNS tube (2,5 ml)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intensive care unit: This group will be composed of patients admitted to the intensive care unit who did not receive invasive mechanical ventilation.
- Intensive care unit and invasive mechanical ventilation: This group will be composed of patients admitted to the intensive care unit who did receive invasive mechanical ventilation.

SUMMARY:
The intensive care unit (ICU) is recognizably detrimental to sleep and circadian health, and critical survivors frequently report the presence of alterations in this regard after hospital discharge. However, an appropriate evaluation of sleep and circadian rhythms is often neglected given the high associated cost and/or the need of collaboration of the patients. In this project, the investigators propose alternatives to ultimately improve the management of sleep and circadian health after critical illness. The researchers will evaluate the role of microRNA (miRNAs) expression profile in identifying the compromised sleep and circadian health of critical patients during the ICU stay, in the short (3 months after hospital discharge), and in the long-term (12 months after hospital discharge). Also, models based on machine learning techniques will be developed to predict adverse outcomes in this regard after hospital discharge.

DETAILED DESCRIPTION:
The intensive care unit environment is recognizably detrimental for sleep and circadian rhythms due to a plethora of factors such as the mistimed and excessive use of artificial light, unusual feeding schedules, night-time noise and interruptions, events associated with acute illness, among others. The reported sleep and circadian alterations often persist after hospital discharge, but there is a lack of quantitative data obtained through appropriate tools for the intensive care unit context, with a proper sample size, and comprising the different profiles of critical patients. The investigators will address this, by evaluating the prevalence of sleep and circadian alterations during the intensive care unit stay and after hospital discharge in the short (3-month follow-up) and long term (12-month follow-up). This will indicate the magnitude of the problem to the healthcare professionals. In the sequence, the investigators will evaluate whether the expected alterations in the sleep and circadian rhythms of critical survivors are associated with important factors for their recovery such as quality of life, mental health, respiratory, and immune function. This is especially relevant given that it will indicate possible clinical markers for compromised sleep and circadian health and thereby increase the probability of patients' referral to a sleep unit whenever a marker is observed.

Despite the frequent complaints of sleep and circadian alterations among critical survivors, the evaluation of sleep and circadian health within this context is often neglected due to a high associated cost and/or the need of collaboration of the patients, which is not always possible. This proposal aims to counteract this matter, by identifying sleep and circadian alterations with the use of a non-invasive, feasible, and reliable approach. Accordingly, the investigators propose to identify such alterations by evaluating the levels of miRNAs, small molecules that are easily obtained through blood collection. This has the potential to increase the overlooked evaluations of sleep and circadian rhythms within this context. Furthermore, with a prompt identification of sleep and circadian alterations, appropriate strategies can be implemented, improving the quality of life and recovery of the patients, also preventing the outcomes associated with compromised sleep and circadian health in the long-term. Finally, the investigators propose to predict sleep and circadian alterations by integrating the information available during the intensive care unit stay with the use of informatic techniques. By doing so, the pertinent management will be implemented according to the needs of each patient. A proper follow-up contributes to the prompt identification of problems in this regard and consequent implementation of therapeutic strategies on time, potentiating the benefits of appropriate sleep and circadian health for the recovery and quality of life. It is important to note that such approach has the potential to aid in decreasing the time and cost-associated burden to which the healthcare system is exposed.

For doing all this, critical patients (n = 271) will be recruited during the ICU stay. Sleep and circadian rhythms will be assessed through actigraphy, and blood samples will be collected for miRNAs expression profile determination. Three months after hospital discharge, a clinical evaluation will be performed, followed by the assessment of the quality of life, mental health, and respiratory function. Sleep and circadian rhythms will be investigated through validated questionnaires and 7 consecutive days of actigraphy. Furthermore, blood will be collected for miRNAs expression profile determination and immune function evaluation. The same procedures will be performed 12 months after hospital discharge

The general objective of the study is to improve the management of sleep and circadian health after critical illness.

The specific objectives are:

1. To evaluate the sleep and circadian health of critical patients in three time-points: during the intensive care unit stay, in the short-term (3 months after hospital discharge), and in the long-term (12 months after hospital discharge).
2. To evaluate possible associations between sleep and circadian health and important factors for the recovery of critical survivors such as quality of life, mental health, respiratory, and immune function in the short and long-term.
3. To evaluate the role of miRNAs expression profile in identifying the compromised sleep and circadian health of critical patients during the intensive care unit stay, in the short, and in the long-term.
4. To identify possible biological events underlying the compromised sleep and circadian health of critical patients during the intensive care unit stay, in the short, and in the long-term.
5. To develop models to predict the compromised sleep and circadian health of critical survivors in the short and long-term.
6. To establish a cohort of critical survivors with available information related to sleep and circadian health to further explore this unravelled research field.
7. To validate the findings in an independent cohort outside Europe.

ELIGIBILITY:
Inclusion Criteria:

* Being older than 18 years old.
* Intensive care unit admission.
* Intensive care unit stay ≥7 days.

Exclusion Criteria:

* Transference to another hospital during hospitalization or follow-up.
* Mental or physical disability that could prevent the proposed evaluations.
* Palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical patients admited to the intensive care unit of the Hospital Arnau de Vilanova de Lleida who meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 271 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Sleep efficiency | 12-month follow-up
  The sleep health of critical patients will be evaluated using this parameter, which will be obtained through 7 days of actigraphy at the 3- and 12-month follow-up. Sleep efficiency is defined as the ratio between total sleep time and the time spent in bed. The following cut-offs are used: i) sleep efficiency ≥ 85% (represents good sleep quality), ii) sleep efficiency <85% (represents inappropriate sleep quality).
Circadian function index (CFI) | 12-month follow-up
  The circadian health of critical patients will be evaluated using this parameter, which will be obtained through 7 days of actigraphy at the 3- and 12-month follow-up. The circadian function index is defined as the average of intradaily variability, interdaily stability, and relative amplitude of the rhythm. There are no specific cut-offs for this parameter. The circadian function index values range from 0-1, in which 1 represents an appropriate circadian function.

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Targa Dias Santos, PhD, Principal Investigator — Institut de Recerca Biomèdica de Lleida
Locations (1):
- Hospital Universitari Arnau de Vilanova, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No